CLINICAL TRIAL: NCT03919864
Title: Caregiver Oncology Needs Evaluation Tool (CONNECT): A Technology-Based Intervention to Connect Lung Cancer Caregivers With Supportive Care Resources
Brief Title: Connect Oncology Needs Evaluation Tool
Acronym: CONNECT-LC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Lung Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00054952; WFBCCC 04319 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2019-04-12; First posted 2019-04-18 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Lung Cancer
Keywords: Lung cancer caregivers
MeSH Terms: conditions — Lung Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONNECT Intervention Group (Other): CONNECT includes a multi-component e-tool with the following: (1) a brief educational video that seeks to empower and educate caregivers about the importance of self-care and benefits of supportive care resource use; (2) an assessment of multidimensional supportive care needs (e.g., psychological, behavioral, social, financial, educational, spiritual); (3) a tailored resource list that includes local and national resources corresponding to caregivers needs (Table1); and (4) an optional automated referral to a caregiver navigator to facilitate connection to resources.
  Interventions: Behavioral: CONNECT Intervention
- CONTROL Group (Other): Control arm participants will receive a generic (i.e., not tailored) printed list of hospital, community, and national supportive care resources. Control participants will not receive the educational video, complete the E-tool Preference survey, or have an option for an automated referral to a caregiver navigator
  Interventions: Behavioral: CONTROL Group

INTERVENTIONS:
Behavioral: CONNECT Intervention — Participants will be included in a multi-component e-tool with brief educational videos, an assessment of multidimensional supportive care needs, a tailored resource list and an optional automated referral to a caregiver navigator. Two weeks after baseline participants will receive re-education and an optional referral.
  Arms: CONNECT Intervention Group
Behavioral: CONTROL Group — Participants will receive a generic printed list of hospital, community, and national supportive care resources.
  Arms: CONTROL Group

SUMMARY:
The purpose of this research study is to evaluate a technology-based intervention, Caregiver Oncology Needs Evaluation Tool (CONNECT), which may increase lung cancer caregivers' knowledge about the benefits of supportive care resources, identify their unmet needs, and connect them with supportive care resources. The investigators will also determine their ability to recruit and keep patients and caregivers in the study.

DETAILED DESCRIPTION:
The long-term goal of this program of research is to improve supportive care delivery and lung cancer caregiver and patient well-being through a caregiver delivered intervention, Caregiver Oncology Needs Evaluation Tool (CONNECT). The investigators propose to evaluate a novel technology-based intervention, CONNECT, informed by theory with input from an advisory panel including a lung cancer caregiver and stakeholders. The purpose of CONNECT is to empower and educate caregivers about the benefits of supportive care resources and to systematically identify unmet needs and connect lung cancer caregivers with tailored supportive care resources. CONNECT is designed to be low cost and to capture the various resources offered in different oncology environments to support future adaptation and dissemination for heterogeneous healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

For Caregivers:

* Caregivers must be providing some capacity of informal (unpaid) care for a patient meeting patient eligibility criteria. If a patient unexpectedly becomes deceased during the study period, caregivers will be allowed to continue participation in the assigned study arm and complete study assessments if they wish to.
* Caregivers must be > 18 years of age, as this study is focused on the experience of adult patient-caregiver dyads.

For Patients:

* Patients must have a current diagnosis of limited stage small cell or stage 1-4 nonsmall cell lung cancer.
* Patients must be currently receiving or planning to receive treatment for their cancer at the time of enrollment. For patients receiving surgery, the eligibility timeframe will include 6 weeks following the date of surgery to account for the acute recovery period.
* Patients must be ambulatory and up more than 50% of waking hours, as measured by an ECOG Performance Status rating of level 0, 1, or 2.
* Patients must be > 18 years of age, as this study is focused on the experience of adult patient-caregiver dyads.
* Patients must be receiving some capacity of informal care from a caregiver meeting the above criteria. If the caregiver unexpectedly becomes deceased during the study period, the patient will be un-enrolled from this study as we are evaluating a caregiver-only delivered intervention.

Exclusion Criteria:

For Caregivers:

• Caregivers cannot read/ communicate in English.

For Patients:

* Patients who are post-treatment survivors at the time of study enrollment. For patients receiving surgery only, this includes the period beyond acute recovery (i.e. ≥ 7 weeks post-surgery).
* Caregivers cannot read/ communicate in English.

Eligibility to participate in the study is conditional on participation of both the caregiver and patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Number of Eligible Participants | Approximately 3 months
  The number of eligible participants who agreed to participate in this study
Accrual | Approximately 3 months
  Number of caregivers who agreed to participate divided by the number of months of recruitment.
Retention of Participants | Approximately 3 months
  Number of participants who completed the T2 assessment divided by the number who agreed to participate
Participants Acceptability of the CONNECT Program Survey | Approximately 3 months
  A 10-item survey developed for study to assess how much caregivers liked different aspects of CONNECT.
Acceptability of CONNECT Program Interview | Approximately 3 months
  A 20-minute qualitative interview to explore factors associated with acceptability. During interviews, CONNECT elements will be reviewed and open-ended questions will be used to elicit feedback on functionality, strengths, and weaknesses of the e-tool. Interview recordings will be transcribed verbatim.

OTHER OUTCOMES:
Supportive Care Service Utilization Survey for Caregivers | Baseline to 3 months
  Survey developed for the purpose of this study to query participants about utilization of supportive care services assessed as part of the CONNECT Preferences Survey. Survey instructions will reflect current assessment (T0, T1, T2 - T0 since your loved one's diagnosis and T1 and T2 since using the online CONNECT program). Caregivers will be asked to think about services or resources from any places they may have gone to for supportive care using the T0, T1, T2 timeframe. Rating scales consists of (Yes, I used this, No, I did not need this, No, I wish this had been available to me and I do not know what this is or if is was available).
PROMIS Emotional Distress-Anxiety-Short Form 8a for Caregivers | Baseline to 3 months
  An 8-item instrument that assesses fear, anxious misery, hyperarousal, and somatic symptoms related to arousal; widely used in oncology populations. Response options range from NEVER to ALWAYS.
PROMIS Emotional Distress- Depression Short Form 8a for Caregivers | Baseline to 3 months
  An 8-item instrument that assesses sadness, guilt, self-criticism, worthlessness, loneliness, interpersonal alienation, as well as loss of Interest, meaning, and purpose. Response options range from NEVER to ALWAYS
Caregiver Reaction Assessment (Burden) for Caregivers | Baseline to 3 months
  A 24-item instrument assessing positive and negative aspects of caregiving (esteem, lack of family support, finances, schedule, and health). Rating scale is based on participants' responses that best describe how they currently feel (Strongly disagree to strongly agree).
Caregiver Quality of Life Index-Cancer (CqoL-Canc) for Caregivers | Baseline to 3 months
  A 35-item instrument assessing dimensions of caregiver quality of life (burden, disruptiveness, positive adaptation, financial concerns). Response options are based on how true each statement has been for the caregiver during the PAST WEEK. Options (not at all, a little bit, somewhat, quite a bit or very much).
FAMCARE (Perceived care quality) Questionnaire for Caregivers | Baseline to 3 months
  A 20-item instrument to assess family caregiver satisfaction with information giving, availability of care, physical patient care, and symptom control. Rating scale options are very satisfied to very dissatisfied.
FAMCARE (Perceived care quality) Questionnaire for Participants | Baseline to 3 months
  A 20-item instrument to assess participant satisfaction with information giving, availability of care, physical patient care, and symptom control. Rating scale options are very satisfied to very dissatisfied.
SF-1247 (Mental and physical well-being) Survey for Participants | Baseline to 3 months
  A 12-item instrument measuring physical and mental well-being of the participants (particularly in the past four weeks). Participants will answer from a scale of 1 = excellent to 5 = poor.
Proportion of Unplanned Hospitalizations | Baseline to 3 months
  Survey designed for the purpose of the study to capture patient self-reported unplanned healthcare utilization. Total score will reflect number of unplanned visits to the emergency room, urgent care, or healthcare provider.
Interventionist Notes - E-Tool Preference Survey | Baseline to 3 months
  A 17-item survey consisting of various resources that participants and their caregivers would like more information on and accessibility of these resources. Response options are YES or NO with the option to select multiple options for obtaining access.
MD Anderson Symptom Inventory for Lung Cancer Questionnaire | Baseline to 3 months
  A 16-item instrument to assess lung cancer specific and general symptoms and the impact on daily functioning. Participants will rate the severity of their symptoms in the last 24 hours based on a scale of 0 = not present to 10 - as bad as you can imagine.
Caregiver Risk Scale | Baseline to 3 months
  A 7-item measure to assess caregiver behaviors for managing self-care. This scale consists of questions that can be answered YES or NO.
Caregiver Barriers Survey | Baseline to 3 months
  A 16-item survey developed for the purpose of this study to assess caregiver barriers to accessing supportive care. Response options: Always, very often, sometimes, rarely, never.
Snyder State Hope Scale for Participants | Baseline to 3 months.
  6-item instrument to assess hope of participants. Score on an 8-point Likert scale with anchor scores of 1 (definitely true) to 8 (definitely false). Higher scores reflect greater state of hope.

CONTACTS AND LOCATIONS:
Overall Officials: Chandylen Nightingale, Ph.D, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT03919864/ICF_000.pdf